CLINICAL TRIAL: NCT04935099
Title: The Effects of a Single Dose of Wild Blueberries on Mood and Cognition in Healthy Young Adults: a Randomized, Double-blind, Placebo-controlled, Crossover Study
Brief Title: The Effects of a Single Dose of Wild Blueberries on Mood and Cognition in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Wild Blueberry Association of North America (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 21/09
Record Dates: First submitted 2021-05-27; First posted 2021-06-22 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Mood; Affect; Cognition
Keywords: blueberry; anthocyanins; flavonoids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry/Placebo (Experimental): In this arm, participants will receive the blueberry intervention first, followed by the placebo one week later.
  Interventions: Dietary Supplement: Wild blueberry powder; Dietary Supplement: Placebo powder
- Placebo/Blueberry (Experimental): In this arm, participants will receive the placebo first, followed by the blueberry intervention one week later.
  Interventions: Dietary Supplement: Wild blueberry powder; Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Wild blueberry powder — 22 g freeze-dried wild blueberry (Vaccinium angustifolium) powder, mixed with 250 ml water, and served in an opaque container.
Dietary Supplement: Placebo powder — 22 g placebo powder matched for macronutrients and flavor, mixed with 250 ml water, and served in an opaque container.

SUMMARY:
This study aims to investigate whether consuming a drink containing powdered blueberries (equivalent to 150 g fresh fruit) can improve mood and cognition in healthy young adults. Blood biomarkers of inflammation and neurotransmitter turnover will be analyzed as well as responses to computer-based cognitive tasks designed to measure verbal memory, executive function, and emotional processing.

DETAILED DESCRIPTION:
The present study will examine the psychological effects of a single dose of freeze-dried wild blueberries using a randomized, double-blind, placebo-controlled, counterbalanced, crossover design. A total of 30 healthy young adults will consume two drinks: one containing 22 g blueberry powder and the other containing 22 g matched placebo powder in counterbalanced order one week apart. The investigators will assess changes in transient mood, cognitive-emotional function, and serum biomarkers of inflammation, neuroplasticity, and monoamine metabolism from baseline to 2 hours post-ingestion.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 25 years of age
* Willingness to provide blood samples

Exclusion Criteria:

* Allergy to blueberries or any other Vaccinium species
* Diagnosis or symptoms of anxiety, depression, or other mental health conditions
* Any medically significant condition (e.g. anemia, gastrointestinal disorders, diabetes)
* Use of psychoactive medication or recreational drugs in the last two weeks
* Current use of medication that could interact with the intervention (e.g. antibiotics)
* Obesity or underweight
* Participation in other interventional studies in the last month
* Pregnancy or lactation

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Global transient mood as measured by PANAS-X | baseline
  The Positive and Negative Affect Schedule - Expanded Form (PANAS-X) is a validated, self-rated measure of affective state, encompassing two general dimensions (positive and negative affect). These will be calculated separately by adding the values of the individual items (21 positive and 25 negative items). Thus, the scales will range from 0 to 84 points for positive affect and from 0 to 100 for negative affect, with a higher score indicating greater positive or negative affect. Positive affect will be considered the primary measure.
Global transient mood as measured by PANAS-X | 2 hours post-ingestion
  The Positive and Negative Affect Schedule - Expanded Form (PANAS-X) is a validated, self-rated measure of affective state, encompassing two general dimensions (positive and negative affect). These will be calculated separately by adding the values of the individual items (21 positive and 25 negative items). Thus, the scales will range from 0 to 84 points for positive affect and from 0 to 100 for negative affect, with a higher score indicating greater positive or negative affect. Positive affect will be considered the primary measure
Negative interpretation bias | baseline
  A negative interpretation bias is defined as a tendency to interpret ambiguous information in a consistently threatening or negative manner, thus serving as an objective indicator of affective state. In this task, participants will be asked to categorize facial expressions of anger, happiness, and surprise as either positive or negative. Interpretation bias will be operationalized as the percent of trials in which surprised faces were rated as negative, out of the total number of surprise trials (48 trials).
Negative interpretation bias | 2 hours post-ingestion
  A negative interpretation bias is defined as a tendency to interpret ambiguous information in a consistently threatening or negative manner, thus serving as an objective indicator of affective state. In this task, participants will be asked to categorize facial expressions of anger, happiness, and surprise as either positive or negative. Interpretation bias will be operationalized as the percent of trials in which surprised faces were rated as negative, out of the total number of surprise trials (48 trials).
Cognitive flexibility (accuracy on post-switch trials) | baseline
  A task-switching test will be used to assess cognitive performance when switching between two predictable tasks requiring simple numerical decisions. The main outcome of interest is the average accuracy of responses to post-switch trials (those immediately following a switch to a new task).
Cognitive flexibility (accuracy on post-switch trials) | 2 hours post-ingestion
  A task-switching test will be used to assess cognitive performance when switching between two predictable tasks requiring simple numerical decisions. The main outcome of interest is the average accuracy of responses to post-switch trials (those immediately following a switch to a new task).
Delayed verbal memory on RAVLT | baseline
  The Rey Auditory Verbal Learning Test (RAVLT) is a standard neuropsychological assessment designed to evaluate verbal memory. The participant hears a list of 15 words and is asked to recall as many words as possible. This procedure is repeated five times. The main outcome of interest is the number of correctly recalled words 20 minutes after the last presentation of the list of words (Trial A7).
Delayed verbal memory on RAVLT | 2 hours post-ingestion
  The Rey Auditory Verbal Learning Test (RAVLT) is a standard neuropsychological assessment designed to evaluate verbal memory. The participant hears a list of 15 words and is asked to recall as many words as possible. This procedure is repeated five times. The main outcome of interest is the number of correctly recalled words 20 minutes after the last presentation of the list of words (Trial A7).
Serum brain-derived neurotrophic factor (BDNF) | baseline
  Serum levels of BDNF will be analyzed using enzyme-linked immunosorbent assay (ELISA).
Serum brain-derived neurotrophic factor (BDNF) | 2 hours post-ingestion
  Serum levels of BDNF will be analyzed using enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Distinct affective states as measured by PANAS-X subscales | baseline
  The following affective states will be examined separately as defined by the PANAS-X subscales: Joviality (Happiness), Self-Assurance, Attentiveness, Fatigue, Serenity. Higher scores will indicate greater intensity of the respective affective state.
Distinct affective states as measured by PANAS-X subscales | 2 hours post-ingestion
  The following affective states will be examined separately as defined by the PANAS-X subscales: Joviality (Happiness), Self-Assurance, Attentiveness, Fatigue, Serenity. Higher scores will indicate greater intensity of the respective affective state.
Reaction time to positive stimuli | baseline
  The average reaction time to correctly categorized happy faces in the facial expression task.
Reaction time to positive stimuli | 2 hours post-ingestion
  The average reaction time to correctly categorized happy faces in the facial expression task.
Reaction time to negative stimuli | baseline
  The average reaction time to correctly categorized angry faces in the facial expression task.
Reaction time to negative stimuli | 2 hours post-ingestion
  The average reaction time to correctly categorized angry faces in the facial expression task.
Attentional bias to emotional information | baseline
  Attentional bias to emotional information will be operationalized as the average reaction time to correctly categorized angry faces divided by the average reaction time to correctly categorized happy faces. Thus, a higher value indicates a tendency to attend to and process positive information over negative information.
Attentional bias to emotional information | 2 hours post-ingestion
  Attentional bias to emotional information will be operationalized as the average reaction time to correctly categorized angry faces divided by the average reaction time to correctly categorized happy faces. Thus, a higher value indicates a tendency to attend to and process positive information over negative information.
Cognitive flexibility (accuracy on remaining trials of task-switching test) | baseline
  The average accuracy (in %) of responses to the remaining trials of the task-switching test will be measured as a secondary outcome. In this task, participants have to switch between two predictable tasks requiring simple numerical decisions.
Cognitive flexibility (accuracy on remaining trials of task-switching test) | 2 hours post-ingestion
  The average accuracy (in %) of responses to the remaining trials of the task-switching test will be measured as a secondary outcome. In this task, participants have to switch between two predictable tasks requiring simple numerical decisions.
Choice reaction time (post-switch trials) | baseline
  The average reaction time of correct responses to post-switch trials of the task-switching test.
Choice reaction time (post-switch trials) | 2 hours post-ingestion
  The average reaction time of correct responses to post-switch trials of the task-switching test.
Choice reaction time (remaining trials of task-switching test) | baseline
  The average reaction time of correct responses to remaining trials of the task-switching test.
Choice reaction time (remaining trials of task-switching test) | 2 hours post-ingestion
  The average reaction time of correct responses to remaining trials of the task-switching test.
Final acquisition on RAVLT (Trial 5) | baseline
  The number of correctly retrieved words on Trial 5 (List A) of the Rey Auditory Verbal Learning Test.
Final acquisition on RAVLT (Trial 5) | 2 hours post-ingestion
  The number of correctly retrieved words on Trial 5 (List A) of the Rey Auditory Verbal Learning Test.
Recall of interference list on RAVLT | baseline
  The number of correctly retrieved words from the interference list (List B) of the Rey Auditory Verbal Learning Test.
Recall of interference list on RAVLT | 2 hours post-ingestion
  The number of correctly retrieved words from the interference list (List B) of the Rey Auditory Verbal Learning Test.
Immediate recall on RAVLT | baseline
  The number of correctly recalled words on the Rey Auditory Verbal Learning Test 2 minutes after the final presentation of List A (and following the presentation and recall of List B).
Immediate recall on RAVLT | 2 hours post-ingestion
  The number of correctly recalled words on the Rey Auditory Verbal Learning Test 2 minutes after the final presentation of List A (and following the presentation and recall of List B).
Proactive interference on RAVLT | baseline
  Proactive interference on the Rey Auditory Verbal Learning Test is defined as the number of correctly recalled words from the interference List B divided by the number of correctly recalled words on Trial 1 of List A (B1/A1). A higher score indicates less proactive interference.
Proactive interference on RAVLT | 2 hours post-ingestion
  Proactive interference on the Rey Auditory Verbal Learning Test is defined as the number of correctly recalled words from the interference List B divided by the number of correctly recalled words on Trial 1 of List A (B1/A1). A higher score indicates less proactive interference.
Retroactive interference on RAVLT | baseline
  Retroactive interference on the Rey Auditory Verbal Learning Test is defined as the number of correctly recalled words on Trial 6 of List A (the free recall trial after the interference List B) divided by the number of correctly recalled words on Trial 5 of List A (A6/A5). A higher score indicates less retroactive interference.
Retroactive interference on RAVLT | 2 hours post-ingestion
  Retroactive interference on the Rey Auditory Verbal Learning Test is defined as the number of correctly recalled words on Trial 6 of List A (the free recall trial after the interference List B) divided by the number of correctly recalled words on Trial 5 of List A (A6/A5). A higher score indicates less retroactive interference.
Retention on RAVLT | baseline
  Retention on the Rey Auditory Verbal Learning Test is defined as the number of correctly recalled words on Trial 7 of List A (the delayed recall trial at 20 minutes) divided by the number of correctly retrieved words on Trial 6 of List A (A7/A6). Thus, a higher score indicates a higher retention rate.
Retention on RAVLT | 2 hours post-ingestion
  Retention on the Rey Auditory Verbal Learning Test is defined as the number of correctly recalled words on Trial 7 of List A (the delayed recall trial at 20 minutes) divided by the number of correctly retrieved words on Trial 6 of List A (A7/A6). Thus, a higher score indicates a higher retention rate.
Serum monoamine oxidase B (MAO-B) inhibition | baseline
  The activity of the enzyme MAO-B in serum will be analyzed using a fluorometric assay.
Serum monoamine oxidase B (MAO-B) inhibition | 2 hours post-ingestion
  The activity of the enzyme MAO-B in serum will be analyzed using a fluorometric assay.
Serum 3,4-dihydroxyphenylglycol (DHPG) | baseline
  Serum levels of DHPG will be analyzed using liquid chromatography-mass spectrometry (LS-MS) to indirectly determine monoamine oxidase A (MAO-A) activity.
Serum 3,4-dihydroxyphenylglycol (DHPG) | 2 hours post-ingestion
  Serum levels of DHPG will be analyzed using liquid chromatography-mass spectrometry (LS-MS) to indirectly determine monoamine oxidase A (MAO-A) activity.
Serum interleukin-6 (IL-6) | baseline
  Serum levels of IL-6 will be analyzed using enzyme-linked immunosorbent assay (ELISA) as an indication of systemic inflammation.
Serum interleukin-6 (IL-6) | 2 hours post-ingestion
  Serum levels of IL-6 will be analyzed using enzyme-linked immunosorbent assay (ELISA) as an indication of systemic inflammation.
Serum C-reactive protein (CRP) | baseline
  Serum levels of CRP will be analyzed using enzyme-linked immunosorbent assay (ELISA) as an indication of systemic inflammation.
Serum C-reactive protein (CRP) | 2 hours post-ingestion
  Serum levels of CRP will be analyzed using enzyme-linked immunosorbent assay (ELISA) as an indication of systemic inflammation.

OTHER OUTCOMES:
Recognition memory on RAVLT | baseline
  In the final task of the Rey Auditory Verbal Learning Test, participants need to recognize the 15 words from List A from a list of 50 words. Recognition memory is defined as the number of correctly recognized words out of the total number of words.
Recognition memory on RAVLT | 2 hours post-ingestion
  In the final task of the Rey Auditory Verbal Learning Test, participants need to recognize the 15 words from List A from a list of 50 words. Recognition memory is defined as the number of correctly recognized words out of the total number of words.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Psychology and Clinical Languages, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT04935099/Prot_SAP_000.pdf